CLINICAL TRIAL: NCT03004456
Title: Efficacy of Distraction on Reduction of Procedural Pain Associated With Venipuncture in the Pediatric Post-Transplant Population
Brief Title: Distraction for Reduction of Pain Associated With Venipuncture in the Pediatric Post-Transplant Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Assistant Professor of Pediatrics at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAQ8828
Record Dates: First submitted 2016-12-23; First posted 2016-12-28 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Pain, Procedural; Distress, Procedural; Venipuncture
Keywords: Phlebotomy; Pain; Distress
MeSH Terms: conditions — Pain, Procedural; Pain | interventions — Osteogenesis, Distraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Distraction (Experimental): Patients randomized to the "Distraction" group will be permitted to choose an age appropriate application (e.g. movie, game) which will be held for them during the blood draw.
  Interventions: Other: Distraction
- Standard of care (No Intervention): Patients randomized to the "Standard of Care" group will not be provided with an iPad.

INTERVENTIONS:
Other: Distraction — Distraction will be provided by allowing the patient to will choose an age appropriate application (e.g. movie, game) which will be held for them during the blood draw.
  Other Names: iPad
  Arms: Distraction

SUMMARY:
Children with chronic diseases, particularly those who have received transplantation (e.g. cardiac, renal, or liver) are a population who undergo frequent painful procedures, such as venipuncture multiple times per week. There is currently no standard of care for pain reduction during venipuncture for pediatric patients having blood drawn in phlebotomy as an outpatient. The study aims to determine the efficacy of distraction in reducing procedural pain and distress associated with venipuncture in pediatric post-transplant patients.

DETAILED DESCRIPTION:
Children with chronic illnesses experience frequent painful experiences over extended periods of time, and may develop long-term physiological, psychological and behavioral sequelae including increased sensitivity to pain and higher levels of anxiety before painful procedures. There is strong evidence to show that distraction is effective in reducing children's pain and distress during painful procedures. However, the evidence to support distraction, as well as other methods of pain reduction during venipuncture (i.e. vibration, topical anesthetics, sucrose), has primarily focused on children who are previously well, as those with chronic disease are an understudied population with regards to pain reduction during simple procedures. Children with chronic disease or pathology, particularly those who have received transplantation (e.g. cardiac, renal, liver), are a population who undergo frequent painful procedures, such as venipuncture multiple times per week. There is currently no standard of care for pain reduction during venipuncture for pediatric patients having blood drawn in phlebotomy or in the transplant clinics as an outpatient.

The investigators will conduct a randomized control trial comparing two groups: Distraction versus standard of care (i.e. no distraction). The intervention (distraction) will be administered using an iPad and allowing the child to self-select a developmentally appropriate distraction (e.g. game, movie, music). Participants will be videotaped for approximately 1 minute, starting from the time of the venipuncture. This video will be viewed at a later date by two trained study investigators to assess the patient's pain and distress associated with venipuncture, as measured by the OSBD-r, CHEOPS, and FLACC.

ELIGIBILITY:
Inclusion Criteria:

* History of solid organ transplantation
* Undergoing venipuncture

Exclusion Criteria:

* Blood being drawn from a central line

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Faces Pain Scale - Revised (FPS-R) | 1 minute
  Faces Pain Scale is a self-report measure of pain intensity developed for children. The scale is intended to measure how children feel inside. "0" equals "No pain" and "10" equals "Very much pain."

SECONDARY OUTCOMES:
Observational Scale of Behavioral Distress - revised (OSBD-r) | 1 minute
  OSBD-r is an observational measure of procedural distress. The behaviors assessed in the OSBD-r include cry, scream, restraint, verbal resistance, information seeking, emotional support, verbal pain and flail. Distress behaviors are weighted on a 1-4 point scale to reflect the intensity of distress. The higher scores indicated a greater level of distress.
Faces-Leg- Activity-Cry-Consolability (FLACC) | 1 minute
  FLACC is an observational measure of procedural pain. Categories for scoring include Face, Legs, Activity, Cry, and Consolability. Total points assigned for each category may be from zero to ten. The numeric rating scale may be categorized into no pain, mild pain, moderate pain, and severe pain based on the 0 (representing no pain) -10 (severe pain) self-report scale.
Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) | 1 minute
  CHEOPS is an observational scale for evaluating postoperative pain in young children. It includes six categories of pain behavior, each with 3-4 levels and scores range from 4 points (no pain) to 13 points (the worst pain).

OTHER OUTCOMES:
Time to successful venipuncture | Less than 5 minutes
  Defined as the time from placing of tourniquet to completion of collection of the first tube.
Number of attempts necessary for successful blood draw. | Less than 5 minutes
Satisfaction evaluation | Less than 5 minutes
  Satisfaction of phlebotomists and parents will be assessed by a Likert-type survey administered immediately after the blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Tsze, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No